CLINICAL TRIAL: NCT03629392
Title: Dietary Methionine and Cysteine Restriction in Overweight Human Subjects
Brief Title: Methionine and Cysteine Restriction in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Kathrine Vinknes, Kathrine Vinknes, PhD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 239948-B
Record Dates: First submitted 2018-08-02; First posted 2018-08-14 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Overweight
Keywords: Methionine; Cysteine; Energy metabolism; Sulfur amino acids
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant: The diets are similar except for methionine and cysteine, and it is thought that the participants will not be able to identify their treatment allocation by taste.
  Investigator: Randomization will be carried out by an investigator that is not related to the study. All foods will be pre-packaged and delivered to the participants by an unrelated company.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low met/cys diet (Experimental): Dietary intervention
  Interventions: Behavioral: Low met/cys diet
- Moderate met/cys diet (Experimental): Dietary intervention
  Interventions: Behavioral: Moderate met/cys diet
- High met/cys diet (Active Comparator): Dietary intervention
  Interventions: Behavioral: High met/cys diet

INTERVENTIONS:
Behavioral: Low met/cys diet — Dietary intervention with low contents of methionine and cysteine
  Arms: Low met/cys diet
Behavioral: Moderate met/cys diet — Dietary intervention with moderate contents of methionine and cysteine
  Arms: Moderate met/cys diet
Behavioral: High met/cys diet — Dietary intervention with high contents of methionine and cysteine
  Arms: High met/cys diet

SUMMARY:
The aim of this study is to examine the effect of methionine and cysteine restriction on energy and macronutrient metabolism in overweight human subjects

DETAILED DESCRIPTION:
The sulfur-containing amino acid methionine and its downstream metabolite cysteine has been associated with fat mass in animal studies and human observational studies. Some of the proposed mechanisms include an association with lipogenesis, insulin sensitivity and disrupted energy metabolism.

The overall aim of this project is to evaluate the effects of a diet low in methionine and cysteine on markers of lipids, amino acids, glucose and other biomarkers related to energy metabolism, including transcriptomic and protein expression data from adipose tissue and lymphocytes. Overweight and obese but otherwise healthy volunteers will be randomized to receive a diet either low, moderate or high in methionine and cysteine concentrations for 1 week.

This is a pilot study that may be considered an extension of NCT02647970. In addition to the primary and secondary outcomes we will evaluate the feasibility of the intervention and procedures.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25-35 kg/m2

Exclusion Criteria:

* High physical activity
* Smoking
* Drugs
* Chronic disease
* Pregnancy or breastfeeding

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentrations of amino acids | Baseline, Day 1, Day 3 and Day 7 (final visit)
  Measurement of biomarkers of amino acid metabolism, including plasma concentrations of methionine, cysteine and related metabolites
Change in protein expression activity in tissues | Baseline and day 7 (final visit for adipose tissue, Baseline and day 1, 3 and 7 (final visit) for lymphocytes.
  Measurement of protein expression and activity related to methionine and cysteine metabolism in adipose tissue and lymphocytes.

SECONDARY OUTCOMES:
Change in plasma concentrations of fatty acids | Baseline, Day 1, Day 3 and Day 7 (final visit)
  Measurement of fatty acid content in plasma
Change in plasma activity indices of steaoryl-CoA desaturase | Baseline, Day 1, Day 3 and Day 7 (final visit)
  Calculated based onthe ratio of plasma concentrations of products and precursors
Change in protein expression of steaoryl CoA-desaturase in adipose tissue | Baseline and Day 7 (final visit)
  Measurement of protein expression of steaoryl CoA-desaturase in adipose tissue
Change in protein expression of steaoryl CoA-desaturase in lymphocytes | Baseline, Day 1, Day 3 and Day 7 (final visit)
  Measurement of protein expression of steaoryl CoA-desaturase in lymphocytes
Change in steaoryl CoA-desaturase activity in adipose tissue | Baseline and Day 7 (final visit)
  Measurement of enzyme activity of steaoryl CoA-desaturase in adipose tissue
Diet feasibility | Baseline, Day 1, Day 3 and Day 7 (final visit)
  Diet feasibility will be measured by a self-administered questionnaire
Diet compliance | Baseline, Day 1, Day 3 and Day 7 (final visit)
  Compliance with the diet will be measured by a self-administered questionnaire
Body composition | Baseline and day 7 (final visit)
  Measurement of body composition by bioimpedance and dual X-ray absorptometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Result] Olsen T, Ovrebo B, Haj-Yasein N, Lee S, Svendsen K, Hjorth M, Bastani NE, Norheim F, Drevon CA, Refsum H, Vinknes KJ. Effects of dietary methionine and cysteine restriction on plasma biomarkers, serum fibroblast growth factor 21, and adipose tissue gene expression in women with overweight or obesity: a double-blind randomized controlled pilot study. J Transl Med. 2020 Mar 11;18(1):122. doi: 10.1186/s12967-020-02288-x. PMID 32160926
- [Derived] Elshorbagy A, Bastani NE, Lee-Odegard S, Ovrebo B, Haj-Yasein N, Svendsen K, Turner C, Refsum H, Vinknes KJ, Olsen T. The association of fasting plasma thiol fractions with body fat compartments, biomarker profile, and adipose tissue gene expression. Amino Acids. 2023 Mar;55(3):313-323. doi: 10.1007/s00726-022-03229-2. Epub 2022 Dec 21. PMID 36542145